CLINICAL TRIAL: NCT06960252
Title: A Prospective Study on the Cycle-Length Mapping Using the OPTRELL™ Mapping Catheter in Patients With Non-paroxysmal Atrial Fibrillation
Brief Title: Cycle-Length Mapping in Patients With Non-paroxysmal Atrial Fibrillation
Acronym: CLM in AF
Status: Recruiting | Type: Observational
Sponsor: Ting-Yung Chang (Other Government)
Responsible Party: Sponsor-Investigator, Ting-Yung Chang, Physician, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Other Study IDs: 2025-01-013AC
Record Dates: First submitted 2025-04-22; First posted 2025-05-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- non-paroxysmal AF: non-paroxysmal AF admitted for catheter ablation
  Interventions: Device: OPTRELL™ Mapping Catheter

INTERVENTIONS:
Device: OPTRELL™ Mapping Catheter — PVI plus substrate modification of LA chamber coexisting with low unipolar voltage (< 3.0 mv) or bipolar voltage (< 0.5 mv) in SR and stable (STD < 30), fast AF CL detected by CLM module and OPTRELL™ Mapping Catheter.

SUMMARY:
The critical atrial substrates in maintaining persistent atrial fibrillation might be identified by Cycle-Length Mapping (CLM) module. Based on the results of multicenter study in Cycle-Length Mapping between Taipei Veterans General Hospital (Professor Shih-Ann Chen) and IRCCS San Donato Policlinic (Professor Carlo Pappone), targeted CLM driver-ablation provided significant benefits in terms of arrhythmia freedom in the treatment of persistent AF. These findings support a patient-tailored, mapping-based strategy for individuals affected by non-paroxysmal AF. The new ultra-high density mapping catheter, OPTRELL, will be available soon in Taiwan. Therefore, we proposed that the degree of atrial interstitial fibrosis detected by using both unipolar and bipolar voltage map in sinus rhythm and CLM in AF with OPTRELL™ Mapping Catheter would be further better characterization of the atrial substrate and could be potentially critical targeted in eliminating the sources of AF.

As additional substrate mapping provided benefits compared to PVI alone in patients with persistent AF, we hypothesize that combination of electrophysiological and substrate-guided ablation strategy using CLM module with OPTRELL™ Mapping Catheter could be used to guide radiofrequency ablation in the patient with non-paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent forms, and allow to be followed.
2. Symptomatic AF refractory or intolerant to at least one Class 1 or 3 antiarrhythmic medication.
3. Patients with persistent/permanent AF (sustained beyond seven days, or lasting less than seven days but necessitating pharmacologic or electrical cardioversion). Persistent AF is defined as an AF episode which lasts longer than 7 days, Persistent AF which lasted longer than 12 months will be defined as long standing persistent AF.
4. Patients with age equal or greater than 20 years old regardless of gender.

Exclusion Criteria:

1. The presence of an atrial or ventricular thrombus.
2. Patients who are allergic to or unsuitable for use with the contrast media.
3. Pregnant patients or patients who are unavailable to receive X-ray.
4. Patients with severe renal insufficiency. (Glomerular Filtration Rate [GFR] < 15 mg/dl or under dialysis)
5. Patients had autonomic nervous system disorder (e.g. respiratory apnea).
6. Patients with age less than 20 years old or greater than 90 years old regardless of gender.
7. Contraindications to anticoagulation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-paroxysmal AF
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | 12 months
  The endpoints are recurrence of all atrial arrhythmia, including AF, atrial flutter, and atrial tachycardia, and defined as an episode lasting > 30 seconds, 3 months after the ablation, during follow-up with ambulatory ECG monitoring every 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Outside US, Taiwan